CLINICAL TRIAL: NCT03809533
Title: Transplantation of Kidneys of Hepatitis C (HCV) Seropositive Donors to HCV Seronegative Recipients With Subsequent Therapy With Sofosbuvir/Velpatasvir (Epclusa)
Brief Title: The Use of Hepatitis C Positive Kidneys in Hepatitis C Negative Kidney Transplant Recipients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amit D Tevar, MD (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor-Investigator, Amit D Tevar, MD, Associate Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19100135
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplantation; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HCV seropositive non-viremic (HCV Ab+/NAT-) donor (Experimental): Kidney recipients will be monitored for HCV for one year following transplant. When HCV RNA is detected, the transmission-triggered treatment phase will be initiated.
  Recipients will be treated with 12-week oral course of sofosbuvir/velpatasvir (Epclusa®), a fixed-dose combination of a nucleotide analogue HCV NS5B polymerase inhibitor (sofosbuvir - 400mg) and a NS5A inhibitor (velpatasvir - 100mg).
- HCV seropositive viremic (HCV Ab+/NAT+) donor (Experimental): Starting post-operative day 1, kidney recipients will be treated with 12-week oral course of sofosbuvir/velpatasvir (Epclusa®), a fixed-dose combination of a nucleotide analogue HCV NS5B polymerase inhibitor (sofosbuvir - 400mg) and a NS5A inhibitor (velpatasvir - 100mg).
  Interventions: Drug: sofosbuvir/velpatasvir

INTERVENTIONS:
Drug: sofosbuvir/velpatasvir — 12-week, oral, fixed-dose
  Other Names: Epclusa
  Arms: HCV seropositive viremic (HCV Ab+/NAT+) donor

SUMMARY:
This is an open-label, pilot trial to test the safety and efficacy of transplantation of kidneys from hepatitis C seropositive non-viremic (HCV Ab+/NAT-) and HCV seropositive viremic (HCV Ab+/NAT+) donors to HCV seronegative recipients on the kidney transplant waitlist. Treatment and prophylaxis will be administered using a transmission-triggered approach for the first scenario (HCV Ab+/NAT- donors, arm 1) and a prophylaxis approach for the later scenario (HCV Ab+/NAT+ donors, arm 2).

DETAILED DESCRIPTION:
This is a prospective, single center, pilot, open-label study of transplantation of kidneys of HCVAb+ donors to HCVAb- recipients with subsequent therapy with sofosbuvir/velpatasvir (Epclusa®). Recipients of a kidney from HCVAb+/NAT- donors will be in arm 1 (the transmission-triggered arm) of the study. In this arm, the study will monitor HCV by measuring HCV RNA in renal transplant recipients. If HCV RNA is detected, indicating transmission of HCV, recipients will be treated with sofosbuvir/velpatasvir (Epclusa®) for 12 weeks. Virological response will be assessed at 4 weeks, end of treatment and 12 weeks after completion of therapy.

Recipients of a kidney from HCVAb+/NAT+ donors will be in arm 2 (the prophylaxis arm) of the study. In this arm, patients will be started on a 12-week course of sofosbuvir/velpatasvir (Epclusa®) immediately post-operatively and will undergo close monitoring of HCV RNA for evidence of transmission.

To be eligible for the study, subjects need to be listed for renal transplantation, be not infected with HCV, HBV or HIV, and sign informed consent.

ELIGIBILITY:
Inclusion criteria (recipients):

1. Patients with end-stage renal disease listed for kidney transplantation at UPMC.
2. On chronic hemodialysis or peritoneal dialysis or stage 5 chronic kidney disease (CKD) defined as a glomerular filtration rate < 15 ml/min
3. Age ≥ 18
4. No available living kidney donor
5. Listed for an isolated kidney transplant at UPMC with <60m of accrued transplant waiting time and/or <60m of dialysis time
6. Have panel reactive antibody level of <98%
7. No obvious contraindication to kidney transplant
8. Able to travel to UPMC for routine post-transplant visits and study visits for a minimum of 12 months after transplantation
9. Able to provide informed consent
10. Be willing to use a contraceptive method for a year after transplant

Exclusion criteria (recipients):

1. HIV positive
2. HCVAb or HCV RNA positive
3. Presence of behavioral risk factors for contracting HCV other than being on hemodialysis. These behavioral risk factors are current injection drug use, current intranasal illicit drug use, current percutaneous/parenteral exposures in an unregulated setting.
4. Hepatitis B surface antigen positive
5. History of liver cirrhosis
6. Persistently elevated liver transaminases, defined as ALT/AST at least 3 times the upper limit of normal for a minimum of 3 consecutive months
7. History of atrial fibrillation requiring the use of amiodarone over the past 12m
8. Patients with etiology of renal failure with increased risk of causing early graft failure as assessed by the investigator team
9. Receipt of prior organ transplant
10. Waitlisted for a multi-organ transplant
11. Pregnant women
12. Known allergy to sofosbuvir/velpatasvir
13. Any condition, psychiatric or physical, that in the opinion of the investigator would make it unsafe to proceed with transplantation or interfere with the ability of the subject to participate in the study

Inclusion criteria (donors):

1. HCV antibody positive
2. HCV NAT negative or positive
3. Kidney donor profile index (KDPI) score <85

Exclusion criteria (donors):

1. Confirmed HIV positive (positive HIV-1 antibody, positive HIV-2 antibody, positive p24 antigen and/or positive HIV NAT)
2. Confirmed HBV positive (positive hepatitis B surface antigen and/or HBV NAT)
3. Known ongoing therapy for HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 5 years
  Rate of adverse events due to sofosbuvir/velpatasvir (Epclusa) in patients in each experimental group
HCV free at 1 year | 1 year
  Proportion of participants in each experimental group who are free of HCV at 1 year following transplantation

SECONDARY OUTCOMES:
Transmission rate of HCV from HCVAb+/NAT- donors to HCVAb- recipients | 5 years
Incidence of allograft rejection | 5 years
Incidence of graft loss | 5 years
All-cause mortality | 5 years
Waitlist time after enrollment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Tevar, MD, Principal Investigator — University of Pittsburgh; Fernanda Silviera, MD, Study Director — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual patient data outside of our investigative team. Aggregate data will be shared in publications as appropriate.